CLINICAL TRIAL: NCT00441571
Title: A Phase 1 Study of Radiolabeled Monoclonal Antibody 7E11-C5.3(177Lu-meO-DOTA-7E11;CYT-500) in Patients With Progressive Androgen-Independent Prostate Cancer
Brief Title: Safety Study of a Radiolabeled Antibody (7E11) in Patients With Progressive Hormone Refractory Prostate Cancer
Acronym: CYT-500
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytogen Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 500Lu01
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Metastatic Prostate Cancer
Keywords: prostate cancer; radiolabeled antibody
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 177Lu-CYT-500

SUMMARY:
The proposed phase 1 clinical trial will investigate the safety and tolerability of 177Lu-CYT-500 in patients with metastatic prostate cancer and determine the optimal antibody mass and dose of 177Lu to be used for further study.

DETAILED DESCRIPTION:
The proposed phase I clinical trial will investigate the safety and tolerability of 177Lu-CYT-500 and determine the optimal antibody mass and dose of 177Lu to be used for further study. The biodistribution and pharmacokinetics will also be assessed. Patients with histologically documented prostate cancer that is progressing following castration will be eligible. Two antibody masses will be explored in cohort 1 before dose escalation of the 177Lu begins. If the two antibody masses show no difference in pharmacokinetics or biodistribution, then the lower of the doses will be used. The radiation dose will be escalated in subsequent cohorts. Dose escalation will be permitted when the last patient accrued to the previous cohort has demonstrated count recovery in cycle 1 such that DLT has not been defined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented prostate cancer that is progressing following castration. The disease should not be progressing so as to require palliative treatment within 12 weeks of enrollment based on clinical assessment by the investigator. All patients must have assessable disease by radionuclide and/or radiographic studies.
* Castrate levels of testosterone (<50 ng/ml).
* Karnofsky performance status >60%.
* Patients whose initial hormone treatment (exclusive of neoadjuvant hormone therapy) was a combined androgen blockade approach, e.g. an orchiectomy plus an anti-androgen, or gonadotropin releasing hormone analog and an anti-androgen, must show progression of disease following withdrawal of the anti-androgen prior to enrollment.
* Adequate organ function:

  * Hematologic:

    * ANC >1,500/mm3
    * Platelet count >100,000/mm3
  * Hepatic: Bilirubin <1.5 mg/dL and AST<1.5X's the ULN
  * Renal: Creatinine <1.5 mg/dL or creatinine clearance > 60 mL/min.
  * Coagulation: Prothrombin time < institutional UNL.
* Patients must have recovered from the acute toxicities of any prior therapy, and not received chemotherapy, radiation therapy or other investigational anticancer therapeutic drugs for at least 4 weeks prior to entry into the trial.
* Patients must be at least 18 years of age.
* Subjects will be informed as to the potential risk of procreation while participating in this trial and will be advised to use effective contraception during the entire study period.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the institution.

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III or IV), or severe debilitating pulmonary disease.
* Active CNS or epidural primary tumor or active CNS or epidural metastases.
* An active uncontrolled infection or an infection requiring intravenous antibiotic treatment.
* Participation in another therapeutic clinical trial with an experimental drug, concurrently or within the 4 weeks prior to dosing in this study.
* Lack of recovery from the myelosuppressive effects of prior radiation therapy or chemotherapy.
* Patients who have undergone diagnostic ProstaScint, Myoscint, or Oncoscint scans, or have undergone any other prior administration of a murine protein for diagnostic or therapeutic purposes, without regard to HAMA test results.
* Patients with a history of autoimmune hepatitis or history of autoimmune disease.
* Prior radiation therapy encompassing >25% of the bone marrow
* Prior systemic administration of a therapeutic radiolabeled monoclonal antibody.
* Patients who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse, while taking the drug and for 4 weeks after stopping treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
To investigate the safety and tolerability of treatment with 177Lu-CYT-500 in patients with progressive androgen-independent prostate cancer
To determine the optimal antibody mass and dose of 177Lu-CYT-500 to be used for further study.
To determine the biodistribution and pharmacokinetics of 177Lu-CYT-500

SECONDARY OUTCOMES:
To determine the rate of HAMA induction as a result of treatment with 177Lu-CYT-500

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Morris, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States